CLINICAL TRIAL: NCT02952937
Title: A Randomized, Open-label, Single Dose, Crossover Phase 1 Study to Compare the Pharmacokinetic Characteristics of GLA5PR GLARS-NF1 Tablet 300 mg and GLA5PR GLARS-NF3 Tablet 300 mg in Healthy Volunteers
Brief Title: Bioequivalence Study of Two Formulations of Pregabalin CR(Controlled-release) Table 300 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GLAPR-106
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Neuralgia, Postherpetic; Postherpetic Neuralgia; Diabetic Neuropathies; Diabetic Neuralgia; Diabetic Polyneuropathy; Diabetic Neuropathy, Painful; Neuralgia; Neuropathic Pain; Pregabalin; Pharmacokinetics; Bioequivalent
MeSH Terms: conditions — Neuralgia, Postherpetic; Diabetic Neuropathies; Neuralgia | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): 1. Period 1: GLA5PR GLARS-NF1 tablet 300mg , 1 tab, once a day(QD), after evening meal(Regular Diet), oral administration(PO).
  2. wash-out period: over 7 days.
  3. Period 2: GLA5PR GLARS-NF3 tablet 300mg, 1 tab, once a day(QD), after evening meal(Regular Diet), oral administration(PO).
  Interventions: Drug: GLA5PR GLARS-NF3 tablet 300mg; Drug: GLA5PR GLARS-NF1 tablet 300mg
- Group 2 (Other): 1. Period 1: GLA5PR GLARS-NF3 tablet 300mg , 1 tab, once a day(QD), after evening meal(Regular Diet), oral administration(PO).
  2. wash-out period: over 7 days.
  3. Period 2: GLA5PR GLARS-NF1 tablet 300mg , 1 tab, once a day(QD), after evening meal(Regular Diet), oral administration(PO).
  Interventions: Drug: GLA5PR GLARS-NF3 tablet 300mg; Drug: GLA5PR GLARS-NF1 tablet 300mg

INTERVENTIONS:
Drug: GLA5PR GLARS-NF3 tablet 300mg — A new formulation(3rd.) of Pregabalin CR tablet
  Other Names: Test drug
Drug: GLA5PR GLARS-NF1 tablet 300mg — A new formulation(1st.) of Pregabalin CR tablet
  Other Names: Comparator drug

SUMMARY:
The purpose of this clinical trial is to (1) evaluate the bioequivalence(BE) of GLA5PR GLARS-NF3 tablet 300mg administered regular diet relative to GLA5PR GLARS-NF1 tablet 300mg administered regular diet and (2) determine the safety and tolerability of a single dose of GLA5PR GLARS-NF3 tablet 300mg administered regular diet and GLA5PR GLARS-NF1 tablet 300mg administered regular diet.

DETAILED DESCRIPTION:
To assess the single dose pharmacokinetics, safety, and tolerability of GLA5PR GLARS-NF3 tablet 300mg administered regular diet relative to GLA5PR GLARS-NF1 tablet 300mg administered regular diet. IP will be administered 1 tablet(300mg) once a day(QD) after evening meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who, at the time of screening, are the age of older than 19 years.
* Subjects who have BMI more than 17.5kg/m2 and less than 30.5kg/m2 and body weight more than 55kg.
* There is no congenital disease or within 3 years of chronic diseases.
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead electrocardiogram (ECG) or clinical laboratory tests.
* Subjects who signed and dated the informed consent form(approved by IRB) after understanding fully to hear a detailed explanation in the clinical trial
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* A subject with any history of gastrointestinal disease (e.g., Crohn's disease, acute or chronic pancreatitis, and others) and surgery (except for simple appendectomy or repair of a hernia), which can influence the absorption of investigational products.
* A subject who has the following clinical laboratory test results

  ☞ Liver Function Test (AST, ALT) > three times the upper limit of the normal range
* History of regular alcohol consumption exceeding 210g/week(12g = 125 mL of wine, 10g = 250 mL of beer, 10g = 50 mL of hard liquor) within 6 months of Screening.
* A subject who has participated in any other clinical trials and had medication within 3 months prior to the first administration of investigational product. (The end date of another clinical trial is based on the last day of the administration)
* A subject who has the following vital signs results in sitting position at the time of the screening :

SBP ≤ 90 mmHg or DBP ≤ 60 mmHg.

* A subject with a history of drug abuse or a positive urine drug screening for drug abuse
* A subject who has taken the drugs that induce and suppress drug-metabolizing enzymes within 30 days prior to investigational product administration.
* A smoker who consumes more than 20 cigarettes/days
* A subject who has taken any ethical-the-counter drug or has taken any over-the-counter drug within 10days before the investigational product administration
* A subject who has donated whole blood within 2 months or blood components within 1 month prior to the investigational product administration
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation.
* A subject who is unable to take regular diet during the study period.
* Abnormal diet that may affect absorption, distribution, metabolism and excretion of drugs
* History of sensitivity to pregabalin, gabapentin, or other alpha2 delta ligands.
* Evidence of hereditary disease, including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* A subject who is not eligible for the study due to reasons on the investigators' judgment.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
AUClast of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)
Cmax of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)

SECONDARY OUTCOMES:
AUCinf of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)
Tmax of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)
t1/2 of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)
CL/F of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)
Vd/F of Pregabalin | Immediately pre-dose(0h), post-dose 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36 hr(14 points)

OTHER OUTCOMES:
Adverse events, Vital signs, Physical examinations, Clinical safety laboratories and 12-lead EKG. | Through study completion(Post-study Visit), an average of 1 month
  Post-study Visit: upto 3 ~7 days after last PK sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No